CLINICAL TRIAL: NCT01253733
Title: TAHLC - Texting to Promote Adolescent Health Liaisons and Chronic Disease Management
Brief Title: MD2Me - Texting to Promote Chronic Disease Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huang, Jeannie, M.D. (Individual)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 091146
Record Dates: First submitted 2010-11-30; First posted 2010-12-03 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Cystic Fibrosis; Inflammatory Bowel Disease; Type 1 Diabetes; Chronic Disease Management
Keywords: Cystic Fibrosis; Inflammatory Bowel Disease; Type 1 Diabetes; Chronic Disease Management; SMS; Text messages; Internet; Healthcare Interactions
MeSH Terms: conditions — Cystic Fibrosis; Inflammatory Bowel Diseases; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMS and Internet (Experimental): The SMS and Internet group will receive information, tips, strategies, and questions related to the self management of chronic disease (cystic fibrosis, inflammatory bowel disease, or type 1 diabetes) on a web-based program and via SMS messages.
  Interventions: Behavioral: MD2ME
- Control (No Intervention): The Control group will receive monthly tip sheets on various health topics for adolescents and young adults.

INTERVENTIONS:
Behavioral: MD2ME — The goals of the MD2Me intervention include increasing disease self-efficacy, disease knowledge, and the ability to control one's disease independently. The intervention includes an 8-week web program with weekly behavioral skills, topics on how to navigate the healthcare system, lifestyle tips, a Discussion Board, and text messages.
  Arms: SMS and Internet

SUMMARY:
UCSD researchers are conducting a study aimed to develop and evaluate a chronic disease self management web and text message based program on health-related self-efficacy and frequency of adolescent-conducted healthcare interactions. We hypothesize that users of the program will demonstrate greater gains between baseline and 8 month measures of health related self-efficacy and adolescent-conducted healthcare interactions as compared to the usual care comparison group.

DETAILED DESCRIPTION:
The MD2Me study (or also known as TAHLC), sponsored by the National Institutes of Health is a 2-year randomized controlled trial to develop and test a text message and Internet based intervention among adolescents and young adults with cystic fibrosis, type 1 diabetes, or inflammatory bowel disease. Adolescents and young adults have been a difficult population to engage in healthcare. It is estimated that 1 in 5 adolescents do not get the healthcare they need. Interventions must address how the healthcare system can engage adolescents with chronic disease and provide opportunities to discuss health-related matters and improve disease outcomes.

This study will help fill multiple gaps in the literature by exploring the utility of a push AND pull SMS texting-based application for chronic disease management among youth. Based on social cognitive theory, the intervention will use accessible technology to promote disease management among adolescents with chronic disease as they transition to adult care. The popularity and usage of SMS already demonstrated by adolescents suggests notable promise for the SMS-based TAHLC program to promote chronic disease self-management and healthcare engagement with substantial positive impacts on health among youth with chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* ages 14 - 22 years
* have cystic fibrosis, type 1 diabetes, or inflammatory bowel disease for at least 6 months
* have access to the internet
* speak English
* has a parent that speaks English or Spanish (if primary participant is under 18)
* willingness to attend assessment visits

Exclusion Criteria:

* pregnant or have children
* have a history of substance abuse or other psychiatric disorder that would impair compliance with study protocol

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2009-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Health related self-efficacy | 8 months
  The primary aim of the study will be to develop and test the effect of a texting intervention TAHLC on health-related self-efficacy and frequency of adolescent-conducted healthcare interactions over the study period of 8 months.

SECONDARY OUTCOMES:
Health knowledge | 8 months
  Disease health knowledge
Health literacy | 8 months
  Health literacy
Quality of Life | 8 Months
  Quality of life including depression, self-esteem, and social support will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie Huang, MD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Huang JS, Terrones L, Tompane T, Dillon L, Pian M, Gottschalk M, Norman GJ, Bartholomew LK. Preparing adolescents with chronic disease for transition to adult care: a technology program. Pediatrics. 2014 Jun;133(6):e1639-46. doi: 10.1542/peds.2013-2830. Epub 2014 May 19. PMID 24843066